CLINICAL TRIAL: NCT05275348
Title: Evaluation of Remotely Delivered Versus In-person Enhance Fitness for Arthritis
Brief Title: Delivery of Enhance Fitness Trial
Acronym: DEFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kushang Patel, Research Associate Professor: School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014022; 6 U48DP006398-03-01 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 6U48DP006398 (NIH)
Record Dates: First submitted 2022-02-09; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Arthritis; Rheumatoid Arthritis; Fibromyalgia; Gout; Osteoarthritis; Lupus or SLE
Keywords: physical activity; arthritis; rural
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Fibromyalgia; Gout; Osteoarthritis; Lupus Erythematosus, Systemic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-EF (Experimental): Remote delivery of Enhance Fitness.
  Interventions: Behavioral: Tele-Enhance Fitness
- In-person EF (Active Comparator): In-person delivery of Enhance Fitness.
  Interventions: Behavioral: In-person Enhance Fitness

INTERVENTIONS:
Behavioral: Tele-Enhance Fitness — Tele-Enhance Fitness (tele-EF) is a community-based exercise program for older adults. It is a supervised group exercise program that will meet virtually 3 times a week for 1 hour for 4 months. Each tele-EF class uses a standardized format that includes a 5-minute warm-up phase, 25 minutes of moderate-intensity aerobic conditioning, 20 minutes of progressive strength training, and 10 minutes of cool down involving flexibility and balance exercises. Strength training involves progressive resistance exercises, using adjustable 1- to 10-pound ankle and wrist weights. Tele-EF classes will be led by an instructor trained in administering EF through a virtual format. EF instructors will be able to monitor and correct participant's movements through videoconference. All tele-EF classes are monitored by a "spotter" who watches participants exercise using gallery mode.
  Arms: Tele-EF
Behavioral: In-person Enhance Fitness — Enhance Fitness is a community-based exercise program for older adults. It is a supervised group exercise program that will meet in person 3 times a week for 1 hour for 4 months. Each EF class uses a standardized format that includes a 5-minute warm-up phase, 25 minutes of moderate-intensity aerobic conditioning/walking, 20 minutes of progressive strength training, and 10 minutes of cool down involving flexibility and balance exercises. Strength training involves progressive resistance exercises, using adjustable 1- to 10-pound ankle and wrist weights. Classes will be led by an instructor trained in administering Enhance Fitness.
  Arms: In-person EF

SUMMARY:
Arthritis is a common condition in the United States, and a leading cause of pain and disability. Physical exercise is recommended for managing arthritis, but access to evidence-based exercise programs is limited, particularly in rural areas. Therefore, the investigators propose to evaluate remote delivery of an evidence-based exercise program called Enhance Fitness (EF) that is recommended for arthritis management. The primary purpose of this study is to determine if remotely delivered EF is non-inferior to in-person EF on primary and secondary outcomes.

ELIGIBILITY:
For participants 65 years or older

Inclusion Criteria:

* CDC defined arthritis (answering yes to the following: "Have you EVER been told by a doctor or other health professional that you have some form of arthritis, rheumatoid arthritis, gout, lupus, or fibromyalgia?")
* Community-dwelling
* English-speaking

Exclusion Criteria:

* cognitive impairment (Mini Montreal Cognitive Assessment [Mini MoCA version 2.1] score <11)
* significant, non-corrected visual or hearing impairment
* pregnancy
* physician does not recommend exercise due to a contraindicating health condition

For participants 18-64 years old:

* CDC defined arthritis (answering yes to the following: "Have you EVER been told by a doctor or other health professional that you have some form of arthritis, rheumatoid arthritis, gout, lupus, or fibromyalgia?")
* Community-dwelling
* English-speaking
* One of the following additional criteria: (a) moderate-to-severe functional limitation, (b) low household income, or (c) living in a rural area. The definitions of these additional criteria are shown below.

  1. Functional limitation: Reporting some difficulty or limitation to doing any of the physical activities listed in the PROMIS 10-item Physical Function Short Form (e.g., bathing, dressing, shopping, walking) will be considered to have moderate to severe functional limitation.
  2. Low Income: Given that income and cost of living can vary geographically (e.g., urban vs. rural), the investigators will use the Department of Housing and Urban Development's low income limit that determines eligibility for various housing programs. Low income is 80 percent of the median income for a given household size and location based on the US Census Bureau's American Community Survey. Lookup tables are published online annually. These questions will be asked in the screening questionnaire by the UW Study Team who will then reference the correct lookup tables to check if participant meets the definition for low income.
  3. Rural Area: The investigators will apply the widely used National Center for Health Statistics urban-rural classification scheme to identify rural counties. The UW Study Team will ask potential participants the county that they currently live in during the telephone screening and will reference the National Center for Health Statistics urban-rural codes to check if the county is classified as rural.

Exclusion Criteria:

* cognitive impairment (Mini Montreal Cognitive Assessment [Mini MoCA version 2.1] score <11)
* significant, non-corrected visual or hearing impairment
* pregnancy
* physician does not recommend exercise due to a contraindicating health condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome Measurement Information System (PROMIS) 10-item short form | 6 month follow up
  A 10-item questionnaire that assesses the participant's physical functioning (i.e., one's ability to perform activities that require physical action, such as self-care, walking indoors or outdoors, or climbing stairs).

SECONDARY OUTCOMES:
Pain Interference | Study months: 0, 4, 10, 16
  Measured by the PROMIS 29 Pain Interference Short Form
30-second Sit-to-Stand Test | Study months: 0, 4
  Standard physical test conducted by Enhance Fitness instructors of number of sit to stands in 30 seconds
30-second Bicep Curl Test | Study months: 0, 4
  Standard physical test conducted by Enhance Fitness instructors of number of arm curls in 30 seconds
Timed Up and Go Test | Study months: 0, 4
  Standard physical test conducted by Enhance Fitness instructor of 8 foot timed up-and-go
Depression | Study months: 0, 4, 10, 16
  PROMIS 29 Depression Short Form
UCLA 3-item Loneliness Scale | Study months: 0, 4, 10, 16
  3 question questionnaire used to assess 3 dimensions of loneliness including relational connectedness, social connectedness and self-perceived isolation. Participants rate these domains from 1-3 (hardly ever, some of the time, or often) with a total score from 3-9 with a lower score indicating 'least lonely' and a higher score indicating 'most lonely'.
Fatigue | Study months: 0, 4, 10, 16
  PROMIS 29 Fatigue Short Form
Patient-Reported Outcome Measurement Information System (PROMIS) 10-item short form | Study months: 0, 4, 16
  A 10-item questionnaire that assesses the participant's physical functioning (i.e., one's ability to perform activities that require physical action, such as self-care, walking indoors or outdoors, or climbing stairs).

OTHER OUTCOMES:
International Physical Activity Questionnaire- Short Form | Study months: 0, 4, 10, 16
  Self-reported time spent engaging in types and intensities of physical activity and sitting time.
Exercise Self-Efficacy Scale | Study months: 0, 4, 10, 16
  9 item 0 to 10 scale used to assess participant's confidence in their ability to exercise when presented with obstacles. Total scores range from 0-90 with higher scores indicating higher exercise self-efficacy.
Anxiety | Study months: 0, 4, 10, 16
  PROMIS 29 Anxiety short form
Sleep Disturbance | Study months: 0, 4, 10, 16
  PROMIS 29 Sleep disturbance short form
Ability to Participate in Social Roles and Activities | Study months: 0, 4, 10, 16
  PROMIS 29 Ability to Participate in Social Roles and Activities short form

CONTACTS AND LOCATIONS:
Overall Officials: Kushang V Patel, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States